CLINICAL TRIAL: NCT06746272
Title: Serratus Planus Block After Minimally Invasive Cardiac Surgery: a Prospective Randomized Study
Brief Title: Serratus Planus Block After Minimally Invasive Cardiac Surgery
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Bernhard Zapletal, Anesthesia and Critical care consultant, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1.5; 2020-005220-10 (EudraCT Number)
Record Dates: First submitted 2024-12-14; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Pain, Postoperative
Keywords: analgesia; Serratus Anterior Planus Block; SAPB; pain; minimally invasive; cardiac surgery; MICS
MeSH Terms: conditions — Pain, Postoperative; Agnosia; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SAPB group (Active Comparator): Ultrasound guided Serratus anterior block will be performed according to the analgetic standard in our department.
  Interventions: Procedure: Serratus Anterior Plane Block
- Standard i.v. analgesia group (No Intervention): A sterile plaster will be placed on an appropriate site to blind ICU and PACU personnel of the intervention. Patients will receive i.v. analgesia according to the analgesic standard of care in our department.

INTERVENTIONS:
Procedure: Serratus Anterior Plane Block — Ultrasound guided Serratus anterior block will be performed according to the analgetic standard in our department using an ultrasound guided transducer to inject 2mg/kg of 0.5% ropivacaine with an adjuvant. A sterile plaster will be placed on the puncture site after performing the block. Patients will receive i.v. analgesia according to the analgesic standard of care in our department.
  Arms: SAPB group

SUMMARY:
Many patients receiving MICS (minimally invasive cardiac surgery) suffer from significant postsurgical pain. While systemic analgesic therapy has been proven to be insufficient in a great number of patients, significant unwanted side effects might occur. Therefore, the investigation of peripheral nerve blocks such as SAPB with potential for high benefit and low risk for adverse effects as new treatment options for thoracotomy-pain is relevant. Previous randomized double-blind investigations of this novel technique are lacking. At this moment our department's current standard of care is that, SAPB is performed in patients after MICS in our department if the treating anesthetist is experienced in the procedure and the patient receives i.v. analgesia only without nerve block is he or she is not. If we are able to show a benefit for patients in the SAPB arm, the nerve block may constitute a new standard of care for all MICS patients no only in our department but also after MICS in general.

Patients ≥18 years of age, being treated in the cardiothoracic ICU after elective cardiac surgery performed via lateral minithoracotomy (mitral valve, tricuspid valve, atrial septal defect closure) will be included after signed informed consent before surgery. Allocation concealment is guaranteed by opening of the concealed envelope and performance of the ultrasound guided SAPB or ultrasound only by medical personnel not involved in any of the study procedures.

Randomization will be carried out by a web-based software ('randomizer,). The intervention will be performed after ICU arrival but under sedation and analgesia before extubation to minimize patient discomfort and to ensure double blinding.

Efficacy will be evaluated using Pain Scoring by visual analogue scale (VAS), opioid requirements, postoperative complications, need for rescue analgesia, lung function tests and markers of myocardial stress and inflammatory parameters in the early postoperative period according to our current protocol in the ICU.

DETAILED DESCRIPTION:
As described in the Brief Summary, patients after MICS may suffer from significant post surgical pain, while SAPB is a promising measure for pain relief and avoidance of opioid associated side effects, high quality data after cardiac surgery are lacking.

This singlecenter, prospective, randomized, double-blinded, clinical trial is conducted at the department for cardiothoracic anesthesia of the Medical University of Vienna, Austria, from January 2023. The study is performed in accordance with the Helsinki Declaration. The study protocol was approved by the Institutional Review Board (EC number 1012/2021) and registered at the European Union Clinical Trials Register (EudraCT trial no. 2020-005220-10). Written informed consent will be obtained from all eligible patients before surgery.

Eligibility and exclusion criteria are described in detail under "eligibility". Patients could drop out from the study after surgery (and therefore after randomization, which is performed at the end of surgery) if any criteria preventing early weaning and extubation arise (hemodynamically or respiratory instability or bleeding requiring reoperation).

Patient demographics and baseline characteristics including baseline ling function will be collected preoperatively. After arrival in the ICU intraoperative characteristics including length of surgery and intraoperative analgesia requirements will be collected. Pain will be assessed by ICU nurses blinded to the intervention group using a visual analogue scale (VAS). Assessments (described under "outcome measures" in detail, will be conducted following SAPB or standard intravenous pain therapy, performed according to our department's standards.

SAPB In patients randomized to receive SAPB, the block will be performed during respiratory weaning, while patients are intubated and sedated post-surgery to ensure blinding and prevent patient discomfort. Nursing staff and ICU physicians will leave the room during the block to ensure blinding. After achieving good visual conditions of the latissimus dorsi and the serratus anterior muscles using a 13-6 MHz linear array ultrasound transducer (HFL38xi, Sonosite, WA) in a cephalad-to-caudal direction, a 70-mm 22-gauge needle (USC 70 Evolution, Temena, Germany) will be inserted in plane. After confirming an optimal needle tip position by injecting minimal doses of local anesthetic, interfascial injection of 0.4 ml of ropivacaine 0.5%/kg body weight combined with 0.5 µg/kg patient body weight of dexmedetomidine as an adjuvant to prolong block duration will be performed between the serratus anterior and the intercostal muscles. After SAPB, a sterile dressing will be placed on the Block site to ensure blinding.

Sham intervention/ i.v. analgesia only In patients randomized to receive standard i.v. analgesia, patient preparation will be performed in the same way as in patients randomized to receive SAPB with nursing staff and ICU doctors leaving the room. After sham intervention, a sterile dressing will be placed on the Block site to ensure blinding.

Additionally, piritramide, hydromorphone and remifentanil requirements, as well as rescue non-steroidal anti-inflammatory drug use, will be recorded for up to 48 hours after SAPB or sham intervention. During the same time frame, we will record the level of sedation or agitation using the Richmond Agitation-Sedation Scale (RASS). We will collect data on adverse events after MICS including PONV, pneumothorax, hematoma, local anesthesia toxicity (LAST), delirium, up to the second postoperative day. Routinely measured plasma markers of inflammation and tissue damage, including C-reactive protein (CRP), interleukin 6 (IL-6); procalcitonin (PCT), creatine kinase (CK) and CK-MB are collected up to the second postoperative day, and FEV1 is routinely measured before surgery and 24 and 48 hours after SAPB or sham according to our local protocol. After the second postoperative day, follow-up will continue until hospital discharge, to record LOS in the ICU, LOS in hospital and hospital and 30 day mortality.

The analgesic standard in our department - apart from SAPB - is as follows:

Analgesia during anesthesia: Fentanyl (2-3 µg/kg) is used at induction, with maintenance via fentanyl (150-200 µg/h) or remifentanil (0.2-0.3 µg/kg/min) according to our departmental protocol. Thirty minutes before surgery end, 1000 mg of acetaminophen is administered with 1000mg of metamizole or if contraindicated, 75mg of diclofenac; if remifentanil is used, a piritramide bolus (0.1 mg/kg) is given 10 minutes before discontinuation; with fentanyl, the infusion is tapered and then stopped 15 minutes before planned extubation.

Analgesia after surgery - Following our department's protocol, patients receive metamizole (1000 mg every 8 hours) and hydromorphone (2-4 mg every 12 hours, based on body weight), supplemented with oral hydromorphone (1.3 mg up to 6 times per day) as nurse-controlled analgesia. if rescue doses are exhausted, the basal hydromorphone dose is increased by 20%. Rescue diclofenac is allowed up to twice a day unless contraindicated. Rescue SAPB performed according to the standards above, is allowed from 12 hours after the intervention or later. Rescue analgesia is allowed if VAS despite metamizole and hydromorphone is > or equal to 5.

Patients will be randomly assigned in a 1:1 ratio using an online block randomization list (www.randomizer.at). To maintain blinding, nurses and other physicians will leave the room during the intervention as described above, a sterile dressing will be applied afterwards in both groups. This is to ensure that the treating physicians and ICU nurses are unaware of the assigned group, and patients remain blinded to the intervention throughout the study.

The primary endpoint is average NRS within 12h after SAPB or standard i.v. analgesia respectively secondary endpoints include opioids 12h, 12-24h and 24-48h after SAPB or standard i.v. analgesia respectively. Further secondary endpoints are described under "outcome measures".

Opioid analgesia after SAPB and sham intervention is performed according to the standard above and converted to parenteral opioid equivalents (PME) (https://opimeter.usz.ch). Remifentanil is excluded from PME calculations due to the impracticality of its conversion. Instead, remifentanil use and dose is compared separately between groups.

For sample size planning a standard deviation of 2.6 points is assumed for the primary endpoint, based on previously reported findings (Toscano A. et al. The Serratus Anterior Plane Study: Continuous Deep Serratus Anterior Plane Block for Mitral Valve Surgery Performed in Right Minithoracotomy. J Cardiothor Vasc An 2020;34(11):2975-82.). An interim analysis with the possibility for early stopping for efficacy is planned after 50% of the maximal sample size has been achieved. The study may be concluded at interim if the adjusted one-sided significance levels of 0.001525 are exceeded in order not to withhold an effective treatment from patients in the standard i.v. analgesia group. Adjusted significance levels for the interim and final analyses are calculated using the Lan-DeMets alpha spending function approximating the O'Brien-Fleming boundaries to control the overall type I error rate at one-sided level of 0.025. We calculated that under these assumptions a maximal sample size of 28 patients per group will be required to detect a mean difference of 2.0 points (20% of the range of possible values) using a two-sample t-test with 80% power. To account for up to 15% drop-outs, a maximum sample size of 32 patients per group is planned.

The primary endpoint, average VAS for postoperative pain within the first 12 hours, will be compared between study groups using a two-sample Welch t-test. The primary outcome is as mean of the averaged VAS score over the first 12 hours. Further continuous endpoints presented in figures and tables including VAS scores for individual points up to 48 hours, PME and remifentanil dosages are compared between groups using t-tests and means (SD) or Mann-Whitney U tests and medians [IQR] are calculated for descriptive purposes. Binary secondary endpoints including rescue analgesia with NSAIDs are compared between groups using Chi-squared tests and described by absolute frequencies and proportions. For secondary endpoints, P < 0.05 (two sided) was considered significant, the analysis of secondary endpoints will be regarded as exploratory.

No imputation will be used in patients with incomplete outcome data. Microsoft Excel, IBM SPSS for Windows and Prism are used for data collection in a database, analysis and construction of figures.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or more
* patients undergoing cardiac surgery through a thoracotomy incision
* patients having surgery performed by a Cardiac Surgeon at the Medical University of Vienna
* patients being treated in the 16 bed primary cardiothoracic ICU 13B-HTG at the Medical University of Vienna
* patients being treated in the 4 bed PACU of the cardiothoracic and vascular anesthesia department at the Medical University of Vienna
* signed patient consent prior to surgery

Exclusion Criteria:

* patients requiring full sternotomy or emergency surgery
* Allergy to amid-type local anesthetics
* patients less that 18 years of age at the time of surgery
* patients intubated >48h prior to surgery
* Infection at the site of the Serratus Anterior Plane Block
* Known bleeding diathesis with increased risk of hematoma at the block site
* Known opioid abuse
* Allergy to (metamizole AND acetaminophen) OR (hydromorphone AND Piritramide)
* Active pulmonary infection at the time of surgery
* Patient refusal prior to surgery
* Inability to communicate
* BMI ≥40
* Patients with known dementia or/and a legal guardian for medical issues
* Patients unable to understand the study measures and are not able to complete pain assessment forms.
* Known pregnancy
* Severe cardiorespiratory disturbances such as high respiratory support (>0,7 FiO2 or driving pressure >25mbar) or high catecholamine support (>0,5mcg/kg/min Norepinephrine and/or >5IE Vasopressin/h) making fast track intensive care with extubation in the first 24 hours after arrival in the ICU and ERAS impossible
* Patients with unanticipated prolonged intubation >24h after arrival in the ICU
* Postoperative ECMO support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Score: VAS 0-10 | 12 hours after successful respiratory weaning
  average pain scores (VAS 0-10) reported according to our department's standards immediately after extubation, and if feasible 2, 4, 6,8,10,12 hours after SAPB (or standard i.v. therapy respectively)

SECONDARY OUTCOMES:
postoperative morphine equivalents | 0-12 hours, 12-24 hours, 24-48hours after successful respiratory weaning
  Measurement of opioid requirements (parenteral morphine equivalents) in the early postoperative period (0-12h, 12-24h and 24-48h after SAPB or standard i.v. pain therapy respectively) in the block group compared to the standard i.v. analgesia group. Analgesia in both groups will be administered according to our department's standards.
VAS at 2, 4, 6, 8, 10, 12, 16, 24, 48 hours | 2-48 hours after application of the serratus block (SAPB)
  difference in VAS at 2, 4, 6, 8, 10, 12, 16, 24, 48 hours after application of the serratus block (SAPB) or standard i.v. pain therapy respectively. Analgesia in both groups will be performed according to our department's standards.
complications from the block, surgery or from postoperative pain | 0-48 hours after conclusion of respiratory weaning
  Complications after MICS (clinically significant pneumothorax, PONV, delirium, hematoma, LAST (local anesthesia systemic toxicity)) will be recorded according to our department's standards
pulmonary function | 0-48 hours after conclusion of respiratory weaning
  pulmonary dysfunction by means of preoperative and postoperative FEV1 will be assessed according to our department's standards
inflammation and myocardial stress parameters | immediately postoperatively, on postoperative day 1 and on postoperative day 2 after MICS
  CRP, IL-6, PCT, CK, CK-MB, NT-PRO-BNP measurements after SAPB or standard i.v. pain therapy according to our departmental standards
rescue analgesia | up to postoperative day 2 after MICS
  rescue analgesia by Diclofenac or SAPB according to our department's standards

OTHER OUTCOMES:
LOS in the ICU, LOS in hospital, hospital and 30 day mortality | up tp 30 days after MICS
  length of stay in the ICU, in hospital and hospital and 30 day mortality after surgery will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Zapletal, M.D., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/72/NCT06746272/Prot_SAP_000.pdf